CLINICAL TRIAL: NCT02877589
Title: Interest of Routine Screening for Hepatitis B and C in Patients Receiving Chemotherapy for Solid Tumors
Acronym: HepScreen
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao002
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Hepatitis B Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- solid tumor: Patients receiving chemotherapy for solid tumors in Ambulatory Medicine Unit of the Reims University Hospital (France) between May 14, 2012 and July 31, 2013.
  Interventions: Other: hepatitis B virus (HBV) and hepatitis C virus (HCV) serologies and a screening questionnaire to detect risk factors of hepatitis B virus (HBV) and hepatitis C virus (HCV)

INTERVENTIONS:
Other: hepatitis B virus (HBV) and hepatitis C virus (HCV) serologies and a screening questionnaire to detect risk factors of hepatitis B virus (HBV) and hepatitis C virus (HCV)

SUMMARY:
Immunosuppression induced by cancer treatment increases the risk of hepatitis B virus (HBV) and hepatitis C virus (HCV) reactivations. These viral reactivations may be asymptomatic but can cause fulminant hepatitis and death. More, they impact the treatment of cancer by chemotherapy delays or stops. They can occur during cancer treatment but also after stopping, at the immunological rebound. This risk persists for at least 6 months after cessation.

The key to the prevention, and the first step, is serological testing. It is also the main problem because international recommendations diverge. Hepatologists and infectious disease specialists recommend routine screening HBV of all candidates for immunosuppressive therapy. These recommendations are more implemented by hematologists, given the frequency of HBV reactivation associated to haematological malignancies. Clinical oncology societies guidelines suggest a selective screening in case of risk factors of hepatitis B or in patients with a strong immunosuppression (such as anti-CD20 based treatment, stem cell transplantation or lymphoma treatment).

The consequence of these differences is a sub-screening by oncologists and the persistence of fatal cases. Screening before cytotoxic chemotherapy for solid tumors in countries with low prevalence of HBV and HCV virus is questionable. Selective screening of patients at risk HBV and HCV can be assessed.

DETAILED DESCRIPTION:
The aims of the study were :

evaluate the seroprevalence of hepatitis B virus (HBV) and hepatitis C virus (HCV) in patients receiving cytotoxic chemotherapy for solid tumors.

assess the relevance of screening questions to detect risk factors of hepatitis B virus (HBV) and hepatitis C virus (HCV) and to analyze the patients with superior risk of viral reactivation

ELIGIBILITY:
Inclusion Criteria:

* patients receiving chemotherapy for solid tumors in Ambulatory Medicine Unit of the Reims University Hospital (France) between May 14, 2012 and July 31, 2013

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving chemotherapy for solid tumors in Ambulatory Medicine Unit of the Reims University Hospital (France) between May 14, 2012 and July 31, 2013
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
hepatitis B virus (HBV) serological status | Day 0
  Serological status for hepatitis B virus (HBV) classified in "HBV exposed", "HBV vaccine" and "HBV negative"

SECONDARY OUTCOMES:
hepatitis C virus (HCV) serological status | Day 0
  Serological status for hepatitis C virus (HBC) classified in "HBC positive" and "HBC negative"

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Brasseur M, Heurgue-Berlot A, Barbe C, Brami C, Rey JB, Vella-Boucaud J, Dabouz F, Deslee G, Grange F, Volet J, Bouche O. Prevalence of hepatitis B and C and sensibility of a selective screening questionnaire in patients receiving chemotherapy for solid tumors. BMC Cancer. 2015 Dec 23;15:999. doi: 10.1186/s12885-015-2033-z. PMID 26694960